CLINICAL TRIAL: NCT04806971
Title: Association Between Vitamin D Receptor, Interleukin-1A and Interleukin-1B Gene Polymorphisms and Stage III Grade B/C Periodontitis
Brief Title: Vitamin D Receptor, Interleukin-1A and Interleukin-1B Gene Polymorphisms in Periodontitis
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: SAG-K-170118-0002
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis; Polymorphism, Restriction Fragment Length
Keywords: Vitamin D receptor; Polymorphism; Periodontitis,; Interleukin-1B; Interleukin-1A
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis: Patients with grade B / C, stage III periodontitis were classified based on the new classification criteria.Clinical attachment loss ≥5 mm, probing depth (PD) ≥6 mm, ≥20 teeth and radiographic bone loss extending to the root middle third. Grade was assessed considering the radiographic bone loss in the most affected tooth in the dentition as a function of age (Grade B=0.25-1.0, Grade C= >1.0).
- Healthy: The periodontally healthy subjects without any clinical sign of inflammation,not showing a history of periodontitis; PD ≤3 mm; <10% of sites with BOP; an absence of detectable bone loss and/or attachment ; without extensive caries or restorations and presence of at least 28 permanent teeth. In addition, all the control subjects showed the absence of any local or systemic pathology.

SUMMARY:
Background: The aim of the study is to find out the prevelance of VDR (rs731236), IL1B (rs1143634) and IL1A (rs1800587)gene polymorphisms in Turkish population and their association with stage III grade B / C periodontitis.

Methods: Individuals who were found to be systemically and periodontally healthy (N = 100) after clinical and radiographic examination and who were diagnosed with Stage III Grade B / C periodontitis (N = 100) were included in the study. Gingival index, Plaque index, bleeding on probing, clinical attachment level and pocket depths of the patients were recorded. subjects genotyped for rs731236, rs1143634 and rs1800587 gene polymorphisms with Real Time Polymerase Chain Reaction.

DETAILED DESCRIPTION:
In this study we recruited 200 participants from the Periodontology Clinics. Periodontal clinical parameters such as plaque index, gingival index, probing depth and clinical attachment level were assessed. Genotyping rs731236, rs1800587 and rs1143634 gene polymorphisms was performed by Real Time Polymerase Chain Reaction.Statistical analysis was done by the statistical software package SPSS v16. SNPassoc.

ELIGIBILITY:
Inclusion Criteria:

systemically healthy, previously untreated periodontitis patients

Exclusion Criteria:

presence of systemic disease such as diabetes, rheumatic fever, liver or kidney diseases, neurologic deficiencies, immunologic diseases; pregnancy; smoking; receive of any medication which may affect periodontal tissues; used antibiotics for any purpose within 6 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 200 subjects were recruited from the Marmara University, Faculty of Dentistry, Clinics of Periodontology
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
IL-1A gene polymorphism | baseline
Interleukin-1B gene polymorphism | baseline
Vitamin D Receptor gene polymorphism | baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University, Istanbul, Maltepe
  - Marmara University Dental Faculty Periodontology Department, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided